CLINICAL TRIAL: NCT01448590
Title: Systematic Review: Post Dural Puncture Headache After Accidental Dural Puncture: Does Insertion of Spinal Catheter Decrease Incidence of Headaches?
Brief Title: Post Dural Puncture Headache After Accidental Dural Puncture
Status: Withdrawn | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Lynn Haslam, Nurse Practitioner, Sunnybrook Health Sciences Centre
Other Study IDs: SHSC-Haslam-PDPH
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Post Dural Puncture Headache
Keywords: post dural puncture headache; accidental dural puncture; PDPH; ADP; spinal catheter; epidural catheter; intrathecal catheter; dural puncture; systemic review
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Epidural Resite: After ADP, those patients who receive an epidural resite.
- Spinal catheter: After ADP, those who receive the epidural catheter into the spinal space

SUMMARY:
Epidural anesthesia is associated with potential risks and complications, post dural puncture headache (PDPH) one of the most recognized with epidural or spinal anesthesia. Accidental dural punctures occur with approximately 1.5% of all epidural attempts. Studies have suggested that the use of an intrathecal catheter reduces the incidence of PDPH. A systematic review of the existing literature will identify if there is reliable evidence to support this theory. A secondary outcome, headache severity, will also be explored via incidence rates of epidural blood patch, as this intervention is performed as a treatment for the most severe headaches.

DETAILED DESCRIPTION:
Post dural puncture headache (PDPH) is one of the recognized complications experienced with epidural or spinal anesthesia, resulting from needle puncture of the dura layer of the meninges. This puncture can be deliberate (during spinal anesthesia) or accidental (during epidural anesthesia). Dural punctures allow a leak of cerebrospinal fluid, leading to the characteristic syndrome of PDPH; also known as a spinal headache or low-pressure headache. Accidental dural punctures occur with approximately 1.5% of all epidural attempts. Studies have estimated that, within the obstetrical population, headaches resulting from an inadvertent dural puncture are as high as 50% to 75%.

As the risk of accidental dural punctures (ADP) cannot be eliminated, research has focused on possible interventions that may be taken in order to avoid the onset of a PDPH, eliminate its severity, or treat effects. One of the most common and effective treatments being an epidural blood patch (EBP). More recently, threading the epidural catheter directly into the intrathecal space after the dural puncture has been recognized as a viable option.

ELIGIBILITY:
Inclusion Criteria:

* any comparative methodology, including case-control studies, cohort studies, randomized clinical trials, and chart reviews.
* Insertion of the epidural catheter into the intrathecal space at the level of dural puncture, was compared to resiting an epidural catheter at another level

Exclusion Criteria:

* Any intentional dural punctures (spinal anesthesia) or use of spinal microcatheters were excluded

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Obstetrical population
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of PDPH after epidural resite versus Number of PDPH after insertion of epidural catheter into spinal space | 1 year
  Review of literature that compares two interventions - resiting the epidural or insertion of epidural catheter into spinal space. The Primary outcome measure will be the number of post dural puncture headache events in each group.

SECONDARY OUTCOMES:
What is the incidence of epidural blood patches (EBP)? | 1 year
  Looking at the incidence of EBP in the spinal catheter group, in comparison to the resited epidural group.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Haslam, RN MN/ACNP, Principal Investigator — Sunnybrook Health Sciences Centre, Toronto; Eric Goldszmidt, MD FRCPC, Principal Investigator — Mount Sinai Hospital, Canada